CLINICAL TRIAL: NCT03522662
Title: An Experimental Medicine Study to Characterise the Importance of IL-18 Production and to Evaluate the Therapeutic Potential of IL-18 Blockade With GSK1070806 in Subjects With Behcet's Disease
Brief Title: Anti IL-18 (GSK1070806) in Behcet's Disease
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Dr. Rona Smith, Dr Rona Smith, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Behcet1070806
Record Dates: First submitted 2018-05-01; First posted 2018-05-11 (Actual); Last update posted 2018-05-11 (Actual); Status verified 2018-05

CONDITIONS: Behcet's Disease
MeSH Terms: conditions — Behcet Syndrome | interventions — GSK1070806

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: GSK1070806 — Single 10mg/kg infusion on Day 0
  Other Names: anti IL-18

SUMMARY:
The primary outcome measure of the study is to demonstrate the safety and tolerability of GSK1070806 in the Behcet's disease population at 24 weeks, with biochemical and clinical efficacy and mechanistic studies to further explore the pathogenesis of Behcet's disease important secondary and exploratory outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Have given written informed consent to participate
* Be aged 18 years and over
* Have a diagnosis of Behcet's disease (according to the International Study Group (ISG) diagnostic guidelines or International Criteria for BD (ICBD)).
* Have active disease, severe enough to necessitate the use of biological therapy at the time of enrolment (i.e. Subjects have refractory disease as defined by the UK Centres of Excellence criteria as failure to respond to steroid and/or immunosuppressive therapy with significant or major organ-threatening disease.

Exclusion Criteria:

1. Age under 18 years
2. Allergies to humanized monoclonal antibodies
3. Subjects who have received any of the following agents within 364 days of day 0:

   1. Alemtuzumab
   2. Rituximab or any other B cell depleting or modulating biological agent
4. Subjects who have received any of the following agents within 180 days of day 0:

   1. Cyclophosphamide
   2. Anti-thymocyte globulin
5. Subjects who have received any of the following agents within 90 days of Day 0:

   1. Intravenous immunoglobulin (IVIG)
   2. Plasmapheresis
6. Subjects who have received any of the following agents within 30 days of Day 0:

   1. Anti-TNF (e.g. adalimumab, etanercept, infliximab)
   2. Anti-IL-6 therapy (e.g. tocilizumab)
   3. Interleukin-1 receptor antagonist (e.g. anakinra)
   4. Alpha interferon
   5. Any live vaccine
7. Subjects who have received any other investigational product within 30 days, 5 half lives or twice the duration of the biological effect, whichever is longer.
8. Subjects required more than 15mg prednisolone daily in the 4 week run in phase.
9. Positive human immunodeficiency virus (HIV) antibody test
10. Positive serology for Hepatitis B (HB), defined as: (i) HB surface antigen positive (HBsAg+) OR (ii) HB core antibody positive (HBcAb+)
11. Positive Hepatitis C (HCV) antibody test
12. Evidence of active or latent tuberculosis (TB) as documented by medical history and examination, chest X-rays (posterior anterior and lateral), and a positive (not indeterminate) QuantiFERON®-TB Gold test.
13. Evidence of chronic infection requiring long term antimicrobial therapy
14. Serum IgG level < 3g/l
15. Lymphoma, leukemia, or any malignancy within the past 5 years except for basal cell or squamous epithelial carcinomas of the skin that have been resected with no evidence of metastatic disease for 3 years, and carcinoma in situ of the uterine cervix.
16. QTc interval (single or average) > 480msec or in subjects with bundle branch block QTc > 500msec (these criteria do not apply to subjects with predominantly paced rhythm).
17. Liver function: ALT > 2xULN and bilirubin > 1.5 ULN (isolated bilirubin > 1.5 ULN is acceptable if bilirubin is fractionated and direct bilirubin < 35%)
18. Compliance: is unlikely to comply with scheduled study visits based on investigator judgment or has a history of substance abuse, psychiatric disorder or condition that may compromise communication with the investigator
19. Women who are pregnant or breast feeding
20. Women of child bearing potential who are unwilling or unable to use an acceptable method to avoid pregnancy for one month before and 12 months after administration of GSK1070806

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2018-08-01 (Estimated); Primary Completion 2020-04-01 (Estimated); Study Completion 2020-04-01 (Estimated)

PRIMARY OUTCOMES:
The occurrence of all moderate, severe and life threatening adverse events | 24 weeks
  Events that that are possibly, probably or definitely attributable to a single IV dose of GSK1070806 (10mg/kg)

SECONDARY OUTCOMES:
All adverse events, including mild events | 24 weeks
  Events that that are possibly, probably or definitely attributable to a single IV dose of GSK1070806 (10mg/kg)
Measurement of disease activity | 24 weeks
  Using a clinical scoring tool, the Behcet's disease current activity form (BDCAF)
Measurement of the accumulation of damage | 24 weeks
  Using a clinical scoring tool, the Vasculitis Damage Index (VDI)

OTHER OUTCOMES:
Comparison of serum free IL-18 and total IL-18 levels | 6 weeks
  Pre and post GSK1070806
Comparison of downstream Th1 cytokines | 6 weeks
  Including interferon gamma, IP-10, IL-10, IL-2, IL-1β and TNF. Pre and post GSK1070806.

CONTACTS AND LOCATIONS:
Overall Officials: Rona M Smith, MD MRCP, Principal Investigator — Cambridge University Hospitals NHS Foundation Trust
Locations (1):
- Addenbrooke's Hospital, University of Cambridge NHS Foundation Trust, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No